CLINICAL TRIAL: NCT05765292
Title: Efficacy and Safety of Multi-strain Probiotic on Pancreatic β-cell Function in Type 2 Diabetes Patients
Brief Title: Probiotic Supplementation and Pancreatic β-Cell Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Taras Shevchenko National University of Kyiv (Other); Danylo Halytsky Lviv National Medical University (Other); Kyiv City Clinical Endocrinology Center (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-8
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Type2 Diabetes; Obesity; Insulin Resistance; Obesity, Abdominal
Keywords: probiotics; type 2 diabetes; pancreatic β-cells
MeSH Terms: conditions — Obesity; Insulin Resistance; Obesity, Abdominal; Diabetes Mellitus, Type 2 | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic (Active Comparator): The multiprobiotic which contains of 14 alive probiotic strains of Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic per day.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The multiprobiotic which contains of 14 alive probiotic strains of Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the pa
  Other Names: Symbiter
  Arms: probiotic
Dietary Supplement: Placebo — Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day
  Arms: placebo

SUMMARY:
Probiotics have beneficial effect on obesity related disorders in animal models. Current understanding for the beneficial effects of probiotics in type 2 diabetes strictly relies on animal and clinical data, which mainly focus on their impact on insulin resistance, anthropometric parameters, glycemic control and markers of chronic systemic inflammation. From the other hand, there is a lack of evidence-based probiotic efficacy on pancreatic β-cell function in terms of type 2 diabetes and related metabolic disorders. In this double-blind single center randomized clinical trial, effect of alive multistrain probiotic vs. placebo on pancreatic β-cell function in type 2 diabetes patient will be assessed.

DETAILED DESCRIPTION:
In this single-center double blind, placebo controlled, parallel group study, type 2 diabetes patients from the Kyiv City Clinical Endocrinology Center will be selected. They will be randomly assigned to receive multiprobiotic "Symbiter" or placebo for 8-weeks administered as a sachet formulation in double-blind treatment. Randomization will be done by the study statistician based on a computer-generated list. The groups will be homogeneous according to age, sex and diagnostic criteria. The assignment of groups will be blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.

The multiprobiotic "Symbiter" will be supplied by Scientific and Production Company "O.D. Prolisok". It contains of 14 alive probiotic strains of Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic and placebo per day. All sachets were identical with similar organoleptic characteristics (e.g., taste and appearance).

The pre-randomization period designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients will be instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants will be instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent study will be instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits will be provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy will be compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (aged 18 to 75);
* presence of T2D diagnosis based on the criteria of the American Diabetes Association (plasma glucose in fasting state ≥7.0 mmol/l; plasma glucose at random measuring ≥11.1 mmol/l; HbA1c ≥6.5% or glucose > 11.1 mmol/l 2 hours after tolerance test with 75 g of glucose);
* presence of pancreatic β-cell dysfunction which defined as HOMA2-β<50%;
* treatment with insulin therapy alone or in combination with oral anti-diabetic drugs (metformin and/or sulphonylureas) in a stable dose for at least 3 months prior to randomization;
* HbA1c level 6.5 to 11.0%;
* signed informed consent

Exclusion Criteria:

* presence of T1D;
* intake of anti-diabetic drugs except for those specified in the inclusion criteria (pioglitazone, glucagon-like peptide (GLP-1) analogs, dipeptide-peptidase 4 (DPP-4) inhibitors, etc.);
* severe diabetes-related complications at screening (ie, end-stage diabetic kidney disease, neuropathy requiring pharmacological treatment, proliferative retinopathy, autonomic neuropathy);
* regular intake of probiotics, prebiotics or antibiotics for 3 months prior the inclusion;
* previously diagnosed allergy to probiotics;
* gastrointestinal disorders including food allergy, gluten-sensitive enteropathy, ulcerative colitis;
* an uncontrolled cardiovascular or respiratory disease, an active malignant tumor or chronic infections;
* participant who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated), and/or had a confirmed case of COVID-19 within 4 weeks prior to enrollment;
* participation in another clinical trial;
* pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
β-cell function (%B) | 8 weeks compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
C-peptide | 8 weeks compared to baseline
  C-peptide, ng/ml

SECONDARY OUTCOMES:
HOMA-2IR | 8 weeks compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
insulin sensitivity (%S) | 8 weeks compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
HbA1c | 8 weeks compared to baseline
  HbA1c in %
fasting plasma glucose (FPG) | 8 weeks compared to baseline
  FPG in mmol/L
weight | 8 weeks compared to baseline
  weight in kg
waist circumferences (WC) | 8 weeks compared to baseline
  WC in cm
body mass index (BMI) | 8 weeks compared to baseline
  weight in kg and height in meters will be combined to report BMI in kg/m^2
cytokines levels | 8 weeks compared to baseline
  TNF-α, IL-1β, IL-6, IL-8, INF-γ

CONTACTS AND LOCATIONS:
Overall Officials: Nazarii Kobyliak, Principal Investigator — Bogomolets National Medical University
Locations (4):
- Ukraine (4):
  - Bogomolets National Medical University, Kyiv
  - Kyiv City Clinical Endocrinology Center, Kyiv
  - Taras Shevchenko National University of Kyiv, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savytska M, Kyriienko D, Komisarenko I, Kovalchuk O, Falalyeyeva T, Kobyliak N. Probiotic for Pancreatic beta-Cell Function in Type 2 Diabetes: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial. Diabetes Ther. 2023 Nov;14(11):1915-1931. doi: 10.1007/s13300-023-01474-6. Epub 2023 Sep 15. PMID 37713103